CLINICAL TRIAL: NCT04159025
Title: EBUS-Miniforceps Biopsy Specimen Acquisition for PD-L1 Testing in Nonsmall Cell Lung Cancer: A Feasibility Study
Brief Title: EBUS-Miniforceps Biopsy Specimen Acquisition for PD-L1 Testing in Nonsmall Cell Lung Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: Boston Scientific Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 201910132
Record Dates: First submitted 2019-11-07; First posted 2019-11-12 (Actual); Results first posted 2023-03-01 (Actual); Last update posted 2023-03-01 (Actual); Status verified 2023-02

CONDITIONS: Non Small Cell Lung Cancer; NSCLC
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Endobronchial ultrasound guided miniforceps biopsy (Experimental): * Standard of care convex-probe endobronchial ultrasound and transbronchial needle aspiration followed by rapid on-site evaluation. If evaluation yields a diagnosis of nonsmall cell lung cancer then EBUS-MFB will be performed.
  * With the EBUS bronchoscope, 6 needle punctures will be made into the targeted lymph node with the 22 gauge aspiration needle. The needle will be removed and the 1mm miniforceps will be passed through the working channel of the EBUS-bronchoscope into the targeted lymph node through the puncture site made using the 22 gauge needle using continuous endobronchial ultrasound guidance. The miniforceps will be used to obtain a core biopsy of the targeted lymph node - 8 core biopsies will be obtained from each targeted lymph node using this technique
  Interventions: Device: CoreDx Pulmonary Mini-Forceps

INTERVENTIONS:
Device: CoreDx Pulmonary Mini-Forceps — Manufactured by Boston Scientific
  Other Names: Endobronchial ultrasound guided mini-forceps

SUMMARY:
The incorporation of PD-L1 testing into clinical practice has progressed at a rapid pace, and now offers an additional line of therapy for eligible patients with nonsmall cell lung cancer. The assay used to detect circulating levels of PD-L1 currently requires core biopsies, and is not approved to be used for specimens collected through a needle based cytological technique. Though endobronchial ultrasound guided transbronchial needle aspiration (EBUS-TBNA) has markedly improved the manner in which patients are diagnosed and staged for lung cancer, alternative means of tissue collection may be mandatory to offer patients access to newer lines of therapy such as PD-L1 inhibition. EBUS-miniforceps biopsy may allow bronchoscopists to obtain core biopsy specimens through the technique of endobronchial ultrasound, so that more invasive approaches such as surgery may be avoided. Feasibility using this approach would indicate that all patients being staged with endobronchial ultrasound procedures would be candidates for PD-L1 testing and potential therapy.

This study is proposed to evaluate the feasibility of using endobronchial ultrasound guided miniforceps biopsy (EBUS-MFB) to acquire tissue that is adequate for PD-L1 testing. Feasibility in this study is defined as the ability to obtain adequate material during EBUS procedures to perform PD-L1 testing.

ELIGIBILITY:
Inclusion Criteria:

* Patients with central lung lesion 1cm in size or larger identified on chest CT with the intention to undergo bronchoscopic evaluation and biopsy. The decision to pursue biopsy will be made by the treating physician and agreed upon by the patient.
* Are at least 18 years old
* Are able to provide informed consent
* Are not pregnant as confirmed by bHCG testing prior to procedure

Exclusion Criteria:

* Patients who refuse to participate
* Are less than 18 years of age
* Are pregnant
* Are physically unable to tolerate flexible bronchoscopy or moderate sedation as determined by the bronchoscopist
* Are unable to provide informed consent
* Are on anticoagulant medications and who cannot safely discontinue their medication prior to their procedure at the recommendation of their treating physician

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2020-01-08 (Actual); Primary Completion 2022-02-24 (Actual); Study Completion 2022-02-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alexander Chen, M.D., Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Endobronchial Ultrasound Guided Miniforceps Biopsy
Started | 20
Completed | 20
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Endobronchial Ultrasound Guided Miniforceps Biopsy
Number analyzed (Participants) | 20
Age, Continuous [Median (Full Range); unit: years] | 67 [53 to 84]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 13
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 20
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 4
  White | 16
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 20

OUTCOME MEASURES:

1. Primary Outcome: Feasibility of Utilizing Endobronchial Ultrasound Guided Miniforceps as Assessed by the Number of Participants From Whom Adequate Amounts of Tissue to Perform PD-L1 Testing Was Acquired
Description: * Adequacy will be defined as sufficient core biopsy material to perform the PD-L1 assay specific for nivolumab
  * Any specimen in which the requested assay returns as "insufficient material to perform testing" will be deemed an "inadequate" specimen.
  * Feasibility cannot be determined until the completion of biopsy for all patients enrolled
Time Frame: Completion of biopsy (day 1)
Measure: Count of Participants; unit: Participants
Arm/Group | Endobronchial Ultrasound Guided Miniforceps Biopsy
Number analyzed (Participants) | 20
Participants | 13

2. Secondary Outcome: Rate of Adverse Events
Time Frame: Through 24 hours after biopsy procedure
Measure: Count of Participants; unit: Participants
Arm/Group | Endobronchial Ultrasound Guided Miniforceps Biopsy
Number analyzed (Participants) | 20
Participants | 0

ADVERSE EVENTS:
Time Frame: Adverse events were followed 24 hours post-procedure.
Arm/Group | Endobronchial Ultrasound Guided Miniforceps Biopsy
All-Cause Mortality (participants affected / at risk) | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20
Other Adverse Events (participants affected / at risk) | 0/20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-05-26): https://cdn.clinicaltrials.gov/large-docs/25/NCT04159025/Prot_SAP_000.pdf